CLINICAL TRIAL: NCT02475694
Title: Acute Lung Injury After Cardiac Surgery: Pathogenesis
Acronym: ALI
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Bodil Steen Rasmussen, Professor, PhD, Aalborg University Hospital
Other Study IDs: N-20080016
Record Dates: First submitted 2015-05-21; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Acute Lung Injury; Metabolic Disturbances; Inflammation; Coagulation; Intravascular; Postoperative; Dysfunction Following Cardiac Surgery
MeSH Terms: conditions — Acute Lung Injury; Inflammation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples stored at -80 degrees of Celcius
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — No treatment

SUMMARY:
The purpose of the present study is to visualize the inflammatory response and coagulation disorders during cardiac surgery in order to identify possible predictors for acute lung injury postoperatively.

DETAILED DESCRIPTION:
Acute lung injury after cardiac surgery is a common complication. The pathophysiology is complex and still not fully elucidate. No specific biomarkers are identified and the diagnosis is solely based on impaired oxygenation.

The purpose of the present study is to identify biomarkers of inflammation and coagulation in blood withdrawn simultaneous from the pulmonary artery and the left atrium during surgery and up to 20 hours after weaning from cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* CABG
* In treatment with statins

Exclusion Criteria:

* Acute surgery
* Valve replacement
* In treatment with immunodepressive drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective coronary artery bypass grafting (CABG)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Acute lung injury measured as the fraction of partial pressure of oxygen divided by the fraction of inspired oxygen | Evaluated 72 hours after weaning from cardiopulmonary bypass (CPB)
  Arterial blood gas analysis

SECONDARY OUTCOMES:
Interleukin-1beta | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interleukin-2 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interleukin-4 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interleukin-6 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interleukin-8 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interleukin-10 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Tumor necroting factor-alpha | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Interferon-gamma | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Granulocyte-macrophage colony-stimulating factor | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Measured in blood samples from radial artery, pulmonary artery and left atrium
Thrombin-antithrombin complexes | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB
  Measured in blood samples from pulmonary artery and left atrium
Plasmin-antiplasmin complexes | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB
  Measured in blood samples from pulmonary artery and left atrium
D-dimer | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB
  Measured in blood samples from pulmonary artery and left atrium
Thrombin Fragment 1.2 | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB
  Measured in blood samples from pulmonary artery and left atrium
Metabolomics | The day before surgery; the day of surgery with measurement just before connecting to , immediately after weaning from CPB, 2, 4, 8, 16 and 20 hours after weaning from CPB; and exactly 48 and 72 hours after weaning from CPB
  Metabolomics using the NMR-technique in blood samples from radial artery, pulmonary artery and left atrium

CONTACTS AND LOCATIONS:
Overall Officials: Bodil S Rasmussen, MD, PhD, Principal Investigator — Aalborg University Hospital